CLINICAL TRIAL: NCT01147458
Title: A Phase 2 Randomized, Double-Blinded, Double-Dummy, Placebo And Active Controlled Two Cohort Two-Way Cross-Over, Multi-Centre Clinical Trial To Examine The Pain Relief Produced By 2 Weeks Of Daily Oral Administration Of A 5-Lipoxygenase (5-Lox) Inhibitor PF-04191834 Alone And In Combination With Naproxen In Patients With Flare-Enriched Osteoarthritis Of The Knee
Brief Title: A Study Of The Safety And Efficacy Of PF-04191834 In Patients With Osteoarthritis Of The Knee
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B0041007
Record Dates: First submitted 2010-06-16; First posted 2010-06-22 (Estimated); Results first posted 2013-05-21 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-05

CONDITIONS: Osteoarthritis, Knee
Keywords: Cross-over; safety; efficacy; tolerability; osteoarthritis; knee; pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- PF-04191834 followed by placebo (Experimental): PF-04191834 600 mg BID dose followed by matched placebo plus naproxen placebo.
  Interventions: Drug: PF-04191834; Drug: PF-04191834 placebo; Drug: Naproxen placebo
- Placebo followed by PF-04191834 (Experimental): Placebo followed by 600 mg BID dose of PF-04191834 plus naproxen placebo.
  Interventions: Drug: PF-04191834 placebo; Drug: PF-04191834; Drug: Naproxen placebo
- PF-04191834+Naproxen followed by Naproxen (Experimental): PF-04191834 600 mg BID + Naproxen 500 mg BID followed by Naproxen 500 mg BID plus PF-04191834 placebo
  Interventions: Drug: PF-04191834; Drug: Naproxen; Drug: PF-04191834 placebo
- Naproxen followed by PF-04191834+Naproxen (Experimental): Naproxen 500 mg BID followed by PF-04191834 600 mg BID + Naproxen 500 mg BID
  Interventions: Drug: Naproxen; Drug: PF-04191834 placebo; Drug: PF-04191834

INTERVENTIONS:
Drug: PF-04191834 — 100 mg tablets of PF-04191834 to provide a 600 mg BID dose administered for two weeks
  Arms: PF-04191834 followed by placebo
Drug: PF-04191834 placebo — Matching PF-04191834 placebo tablets to be administered BID for two weeks
  Arms: PF-04191834 followed by placebo
Drug: Naproxen placebo — Matching naproxen placebo tablets to be administered BID for 4 weeks
  Arms: PF-04191834 followed by placebo
Drug: PF-04191834 placebo — Matching PF-04191834 placebo tablets to be administered BID for two weeks
  Arms: Placebo followed by PF-04191834
Drug: PF-04191834 — 100 mg tablets of PF-04191834 to provide a 600 mg BID dose administered for two weeks
  Arms: Placebo followed by PF-04191834
Drug: Naproxen placebo — Matching naproxen placebo tablets to be administered BID for 4 weeks
  Arms: Placebo followed by PF-04191834
Drug: PF-04191834 — 100 mg tablets of PF-04191834 to provide a 600 mg BID dose administered for two weeks
  Arms: PF-04191834+Naproxen followed by Naproxen
Drug: Naproxen — Naproxen 500 mg tablet administered BID for a total of four weeks
  Arms: PF-04191834+Naproxen followed by Naproxen
Drug: PF-04191834 placebo — Matching PF-04191834 placebo tablets to be administered BID for two weeks
  Arms: PF-04191834+Naproxen followed by Naproxen
Drug: Naproxen — Naproxen 500 mg tablet administered BID for a total of four weeks
  Arms: Naproxen followed by PF-04191834+Naproxen
Drug: PF-04191834 placebo — Matching PF-04191834 placebo tablets to be administered BID for two weeks
  Arms: Naproxen followed by PF-04191834+Naproxen
Drug: PF-04191834 — 100 mg tablets of PF-04191834 to provide a 600 mg BID dose administered for two weeks
  Arms: Naproxen followed by PF-04191834+Naproxen

SUMMARY:
PF-04191834 works in animal models by inhibiting one of the enzymes, 5-lipoxygenasein which is involved in the pathway that causes inflammation and pain. The purpose of this study is to test how effective, safe and tolerated PF-04191834 is in patients with osteoarthritis of the knee by itself or with naproxen, particularly to test if patients have less pain.

DETAILED DESCRIPTION:
This study has been terminated in response to a reported serious adverse event (SAE). The sponsor's assessment of the limited data available at the time of the initial SAE report was that the SAE may alter the potential benefit - risk profile of the study medication.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosis of osteoarthritis based on the American College of Rheumatology criteria confirmed by an X-ray
* Subjects must be willing and able to stop all current pain therapy for the duration of the study
* Subjects must be willing and able to complete a daily diary

Exclusion Criteria:

* BMI of >39 kg/m2
* Known allergy or hypersensitivity to naproxen
* Any condition or medical history that might interfere with the subject's ability to complete the study visits and assessments

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2010-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (28):
- United States (23):
  - Pfizer Investigational Site, Peoria, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Carmichael, California
  - Pfizer Investigational Site, Fair Oaks, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Pensacola, Florida
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, South Bend, Indiana
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Edina, Minnesota
  - Pfizer Investigational Site, Saint Paul, Minnesota
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Monroe, North Carolina
  - Pfizer Investigational Site, Fargo, North Dakota
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Arlington, Virginia
- Canada (3):
  - Pfizer Investigational Site, St. John's, Newfoundland and Labrador
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
- Sweden (2):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Stockholm

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0041007&StudyName=A%20Study%20Of%20The%20Safety%20And%20Efficacy%20Of%20PF-04191834%20In%20Patients%20With%20Osteoarthritis%20Of%20The%20Knee

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-04191834 Followed by Placebo: PF-04191834 600 milligrams (mg) twice daily (BID) plus naproxen placebo for 2 weeks with a 2-week washout period, followed by PF-04191834 placebo plus naproxen placebo for another 2 weeks.
- Placebo Followed by PF-04191834: PF-04191834 placebo plus naproxen placebo for 2 weeks with a 2-week washout period, followed by PF-04191834 600 mg BID plus naproxen placebo for another 2 weeks.
- PF-04191834 + Naproxen Followed by Naproxen: PF-04191834 600 mg BID plus naproxen 500 mg BID for 2 weeks with a 2-week washout period, followed by naproxen 500 mg BID plus PF-04191834 placebo for another 2 weeks.
- Naproxen Followed by PF-04191834 + Naproxen: Naproxen 500 mg BID plus PF-04191834 placebo for 2 weeks with a 2-week washout period, followed by PF-04191834 600 mg BID plus naproxen 500 mg BID for another 2 weeks.
Period: First Intervention
Arm/Group | PF-04191834 Followed by Placebo | Placebo Followed by PF-04191834 | PF-04191834 + Naproxen Followed by Naproxen | Naproxen Followed by PF-04191834 + Naproxen
Started | 48 | 47 | 47 | 48
Completed | 34 | 31 | 35 | 34
Not Completed | 14 | 16 | 12 | 14
Not completed — Study terminated by sponsor | 8 | 8 | 7 | 8
Not completed — Protocol Violation | 2 | 3 | 2 | 3
Not completed — Withdrawal by Subject | 3 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 3 | 2 | 3
Not completed — Other | 1 | 2 | 0 | 0
Period: Washout Period of 2 Weeks
Arm/Group | PF-04191834 Followed by Placebo | Placebo Followed by PF-04191834 | PF-04191834 + Naproxen Followed by Naproxen | Naproxen Followed by PF-04191834 + Naproxen
Started | 34 | 31 | 35 | 34
Completed | 34 | 31 | 35 | 34
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | PF-04191834 Followed by Placebo | Placebo Followed by PF-04191834 | PF-04191834 + Naproxen Followed by Naproxen | Naproxen Followed by PF-04191834 + Naproxen
Started | 34 | 31 | 35 | 34
Completed | 25 | 24 | 27 | 30
Not Completed | 9 | 7 | 8 | 4
Not completed — Study terminated by sponsor | 7 | 5 | 5 | 3
Not completed — Protocol Violation | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 1 | 1
Not completed — Other | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive PF-04191834 first, placebo first, PF-04191834 plus naproxen first, and naproxen first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 190
Age Continuous [Mean (Standard Deviation); unit: Years] | 59.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 80

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Western Ontario & McMaster (WOMAC) Osteoarthritis Index Pain Score at the End of Treatment Period 1
Description: The WOMAC Pain subscale, comprised of 5 questions regarding the amount of pain experienced in the index joint, was calculated as the mean of the scores from the 5 individual questions. The WOMAC Pain subscale scores for each question range from 0 to 4 giving a possible overall score range of 0-20, with higher scores indicating higher pain.
Time Frame: Baseline (Day 1 of Visit 3) and end of treatment Period 1 (Day 15+1 of Visit 5)
Population: Full Analysis Set (FAS): included all participants randomized who received at least one dose of study drug, regardless of whether they had efficacy data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-04191834 Followed by Placebo | Placebo Followed by PF-04191834 | PF-04191834 + Naproxen Followed by Naproxen | Naproxen Followed by PF-04191834 + Naproxen
Number analyzed (Participants) | 48 | 47 | 47 | 48
Units on a scale
  Baseline | 11.3 (2.34) | 11.5 (2.81) | 10.8 (2.60) | 11.1 (2.93)
  Change from Baseline | -1.2 (2.49) | -1.6 (3.10) | -1.9 (2.97) | -1.6 (2.93)
Statistical Analysis 1: Comparison: PF-04191834 Followed by Placebo vs Placebo Followed by PF-04191834; The analysis was a mixed model with random participant effect, period and treatment as fixed effects, utilizing the baseline scores (one for each treatment period) as inter- and intra- participant covariates; Test type: Superiority or Other; p = 0.067, ANCOVA; Mean Difference (Net) = 0.56, 80% CI 2-sided [0.08 to 1.04], Standard Error of Mean 0.374
Statistical Analysis 2: Comparison: PF-04191834 + Naproxen Followed by Naproxen vs Naproxen Followed by PF-04191834 + Naproxen; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.701, ANCOVA; Mean Difference (Net) = -0.20, 80% CI 2-sided [-0.67 to 0.28], Standard Error of Mean 0.369

2. Primary Outcome: Change From Baseline in Western Ontario & McMaster (WOMAC) Osteoarthritis Index Pain Score at the End of Treatment Period 2
Description: as for outcome 1
Time Frame: Baseline (Day 28 of Visit 7) and end of treatment Period 2 (Day 43+1 of Visit 9)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-04191834 Followed by Placebo | Placebo Followed by PF-04191834 | PF-04191834 + Naproxen Followed by Naproxen | Naproxen Followed by PF-04191834 + Naproxen
Number analyzed (Participants) | 48 | 47 | 47 | 48
Units on a scale
  Baseline | 9.7 (3.53) | 8.6 (3.15) | 9.7 (2.74) | 10.2 (3.47)
  Change from Baseline | -1.8 (2.58) | -0.6 (2.44) | -1.5 (3.64) | -2.1 (3.03)
Statistical Analysis 1: Comparison: PF-04191834 Followed by Placebo vs Placebo Followed by PF-04191834; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.067, ANCOVA; Mean Difference (Net) = 0.56, 80% CI 2-sided [0.08 to 1.04], Standard Error of Mean 0.374
Statistical Analysis 2: Comparison: PF-04191834 + Naproxen Followed by Naproxen vs Naproxen Followed by PF-04191834 + Naproxen; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.701, ANCOVA; Mean Difference (Net) = -0.20, 80% CI 2-sided [-0.67 to 0.28], Standard Error of Mean 0.369

3. Secondary Outcome: WOMAC Stiffness Domain Score
Description: The WOMAC Stiffness subscale, comprised of 2 questions regarding the amount of stiffness experienced in the index joint, was calculated as the mean of the scores from the 2 individual questions. The WOMAC Stiffness subscale scores for each question range from 0 to 4 giving a possible overall score range of 0-8, with higher scores indicating more stiffness.
Time Frame: Baseline (Day 1 of Visit 3 for Period 1 and Day 28 of Visit 7 for Period 2), Day 15+1 of Visit 5 for Period 1, and Day 43+1 of Visit 9 for Period 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-04191834 Followed by Placebo | Placebo Followed by PF-04191834 | PF-04191834 + Naproxen Followed by Naproxen | Naproxen Followed by PF-04191834 + Naproxen
Number analyzed (Participants) | 48 | 47 | 47 | 48
Units on a scale
  Period 1 Baseline | 4.8 (1.20) | 5.0 (1.41) | 4.7 (1.42) | 4.8 (1.47)
  Period 1 End of Treatment | 4.4 (1.28) | 4.4 (1.44) | 3.8 (1.36) | 4.0 (1.55)
  Period 2 Baseline | 4.2 (1.51) | 3.9 (1.33) | 3.9 (1.44) | 4.4 (1.41)
  Period 2 End of Treatment | 3.3 (1.65) | 3.5 (1.38) | 2.9 (1.31) | 3.6 (1.74)
Statistical Analysis 1: Comparison: PF-04191834 Followed by Placebo vs Placebo Followed by PF-04191834; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = 0.07, 80% CI 2-sided [-0.15 to 0.29], Standard Error of Mean 0.172
Statistical Analysis 2: Comparison: PF-04191834 + Naproxen Followed by Naproxen vs Naproxen Followed by PF-04191834 + Naproxen; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = 0.13, 80% CI 2-sided [-0.09 to 0.35], Standard Error of Mean 0.170

4. Secondary Outcome: WOMAC Physical Function Domain Score
Description: The WOMAC Physical Function subscale refers to the participant's ability to move around and perform usual activities of daily living. The WOMAC Physical Function subscale, comprised of 17 questions regarding the degree of difficulty experienced in the index joint, was calculated as the mean of the scores from the 17 individual questions. The WOMAC Physical Function subscale scores for each question range from 0 to 4 giving a possible overall score range of 0-68, with higher scores indicating worse function.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-04191834 Followed by Placebo | Placebo Followed by PF-04191834 | PF-04191834 + Naproxen Followed by Naproxen | Naproxen Followed by PF-04191834 + Naproxen
Number analyzed (Participants) | 48 | 47 | 47 | 48
Units on a scale
  Period 1 Baseline | 37.7 (9.39) | 39.7 (10.27) | 37.4 (8.50) | 38.7 (10.43)
  Period 1 End of Treatment | 35.4 (9.60) | 35.7 (10.01) | 30.8 (11.30) | 32.0 (13.43)
  Period 2 Baseline | 32.6 (12.37) | 31.6 (9.64) | 31.6 (10.70) | 35.6 (11.46)
  Period 2 End of Treatment | 27.9 (13.11) | 30.8 (11.02) | 25.0 (10.75) | 28.7 (14.95)
Statistical Analysis 1: Comparison: PF-04191834 Followed by Placebo vs Placebo Followed by PF-04191834; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = 1.26, 80% CI 2-sided [-0.34 to 2.85], Standard Error of Mean 1.239
Statistical Analysis 2: Comparison: PF-04191834 + Naproxen Followed by Naproxen vs Naproxen Followed by PF-04191834 + Naproxen; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = -0.34, 80% CI 2-sided [-1.95 to 1.28], Standard Error of Mean 1.252

5. Secondary Outcome: WOMAC Total Score
Description: The WOMAC total score was calculated as the sum of Pain subscale score (5 questions), Stiffness subscale score (2 questions) and Physical Function subscale score (17 questions), with a total of 24 questions(score range:0=none, 4=extreme) giving a possible total score range from 0 to 96 . lower subscale scores represent less pain, less stiffness, or better physical performance.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-04191834 Followed by Placebo | Placebo Followed by PF-04191834 | PF-04191834 + Naproxen Followed by Naproxen | Naproxen Followed by PF-04191834 + Naproxen
Number analyzed (Participants) | 48 | 47 | 47 | 48
Units on a scale
  Period 1 Baseline | 53.7 (11.96) | 56.0 (13.49) | 52.9 (11.57) | 54.8 (14.05)
  Period 1 End of Treatment | 50.0 (12.60) | 49.9 (14.16) | 43.5 (14.96) | 45.4 (18.54)
  Period 2 Baseline | 46.4 (16.94) | 44.2 (13.62) | 45.1 (14.37) | 50.3 (15.96)
  Period 2 End of Treatment | 39.4 (18.13) | 42.6 (15.73) | 35.4 (14.32) | 40.6 (20.99)
Statistical Analysis 1: Comparison: PF-04191834 Followed by Placebo vs Placebo Followed by PF-04191834; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = 2.06, 80% CI 2-sided [-0.13 to 4.25], Standard Error of Mean 1.699
Statistical Analysis 2: Comparison: PF-04191834 + Naproxen Followed by Naproxen vs Naproxen Followed by PF-04191834 + Naproxen; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = -0.33, 80% CI 2-sided [-2.53 to 1.88], Standard Error of Mean 1.709

6. Secondary Outcome: Importance Weighted Total WOMAC Score
Description: Importance weighted total WOMAC score was calculated using all subscales including Pain, Stiffness and Physical Function subscales (24 questions in total,score range: 0=none to 4= extreme,giving a possible overall score range of 0-96).Lower subscale scores represent less pain, less stiffness, or better physical performance.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-04191834 Followed by Placebo | Placebo Followed by PF-04191834 | PF-04191834 + Naproxen Followed by Naproxen | Naproxen Followed by PF-04191834 + Naproxen
Number analyzed (Participants) | 48 | 47 | 47 | 48
Units on a scale
  Period 1 Baseline | 19.7 (4.38) | 20.5 (4.94) | 19.4 (4.26) | 20.1 (5.17)
  Period 1 End of Treatment | 18.3 (4.60) | 18.2 (5.22) | 15.9 (5.51) | 16.6 (6.82)
  Period 2 Baseline | 17.0 (6.23) | 16.2 (5.03) | 16.6 (5.25) | 18.4 (5.88)
  Period 2 End of Treatment | 14.4 (6.65) | 15.6 (5.79) | 13.0 (5.29) | 14.9 (7.71)
Statistical Analysis 1: Comparison: PF-04191834 Followed by Placebo vs Placebo Followed by PF-04191834; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = 0.77, 80% CI 2-sided [-0.03 to 1.58], Standard Error of Mean 0.624
Statistical Analysis 2: Comparison: PF-04191834 + Naproxen Followed by Naproxen vs Naproxen Followed by PF-04191834 + Naproxen; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = -0.16, 80% CI 2-sided [-0.97 to 0.65], Standard Error of Mean 0.628

7. Secondary Outcome: Daily Diary Pain Score During Week 1 of Each Treatment Period
Description: The daily diary pain was assessed using an 11-point numerical rating scale (NRS) ranging from 0 to 10 (0 = no pain; 10 = the worst pain possible).
Time Frame: 4 days prior to baseline visits (Visits 3 for Period 1 and Vist 8 for Period 2) up to 7 days after baseline visits
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-04191834 Followed by Placebo | Placebo Followed by PF-04191834 | PF-04191834 + Naproxen Followed by Naproxen | Naproxen Followed by PF-04191834 + Naproxen
Number analyzed (Participants) | 48 | 47 | 47 | 48
Units on a scale
  Baseline of Period 1 | 6.5 (1.56) | 6.9 (1.36) | 6.4 (1.45) | 6.7 (1.55)
  Week 1 of Period 1 | 6.2 (1.71) | 6.5 (1.52) | 5.4 (1.80) | 5.6 (2.05)
  Baseline of Period 2 | 5.1 (2.18) | 4.8 (2.31) | 5.4 (1.69) | 5.6 (1.85)
  Week 1 of Period 2 | 5.1 (2.27) | 4.8 (2.48) | 4.7 (1.87) | 5.0 (2.04)
Statistical Analysis 1: Comparison: PF-04191834 Followed by Placebo vs Placebo Followed by PF-04191834; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = 0.01, 80% CI 2-sided [-0.18 to 0.20], Standard Error of Mean 0.150
Statistical Analysis 2: Comparison: PF-04191834 + Naproxen Followed by Naproxen vs Naproxen Followed by PF-04191834 + Naproxen; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = 0.12, 80% CI 2-sided [-0.07 to 0.31], Standard Error of Mean 0.147

8. Secondary Outcome: Daily Diary Pain Score During Week 2 of Each Treatment Period
Description: as for outcome 7
Time Frame: Over the last 4 days before baseline visits (Visits 3 for Period 1 and Visit 8 for Period 2) and over the last 6 days before Visit 5 for Period 1 and Visit 9 for Period 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-04191834 Followed by Placebo | Placebo Followed by PF-04191834 | PF-04191834 + Naproxen Followed by Naproxen | Naproxen Followed by PF-04191834 + Naproxen
Number analyzed (Participants) | 48 | 47 | 47 | 48
Units on a scale
  Baseline of Period 1 | 6.5 (1.56) | 6.9 (1.36) | 6.4 (1.45) | 6.7 (1.55)
  Week 2 of Period 1 | 5.8 (1.91) | 5.8 (1.72) | 5.3 (1.66) | 5.6 (2.16)
  Baseline of Period 2 | 5.1 (2.18) | 4.8 (2.31) | 5.4 (1.69) | 5.6 (1.85)
  Week 2 of Period 2 | 4.8 (2.44) | 4.5 (2.58) | 4.4 (1.68) | 4.8 (2.18)
Statistical Analysis 1: Comparison: PF-04191834 Followed by Placebo vs Placebo Followed by PF-04191834; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = 0.09, 80% CI 2-sided [-0.12 to 0.31], Standard Error of Mean 0.168
Statistical Analysis 2: Comparison: PF-04191834 + Naproxen Followed by Naproxen vs Naproxen Followed by PF-04191834 + Naproxen; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = 0.10, 80% CI 2-sided [-0.11 to 0.31], Standard Error of Mean 0.162

9. Secondary Outcome: Rescue Medication Use
Description: Rescue medication use was collected daily in a daily diary, in which participants noted the amount of rescue medication (number of pills) taken each day. Participants were provided with rescue medication paracetamol/acetaminophen throughout the study including the Washout Period and the Initial Pain Assessment Period. Paracetamol/acetaminophen was taken as needed to a maximum of 2000 mg per day, but must be discontinued 48 hours prior to the Baseline visit (Visit 3). From Visit 3 onwards, participants might take up to 2000 mg of paracetamol/acetaminophen per day up to 3 days per week.
Time Frame: Day -7 (Visit 2) up to 28-day follow-up (Visit 10)
Population: Number of subjects analyzed (N) is the number of participants taking rescue mediation.
Measure: Mean (Standard Deviation); unit: Number of pills
Arm/Group | PF-04191834 Followed by Placebo | Placebo Followed by PF-04191834 | PF-04191834 + Naproxen Followed by Naproxen | Naproxen Followed by PF-04191834 + Naproxen
Number analyzed (Participants) | 33 | 30 | 26 | 26
Number of pills
  Period 1 | 1096.1 (310.59) | 1114.5 (367.92) | 1210.2 (442.70) | 1073.7 (409.83)
  Period 2 | 1100.0 (528.15) | 1078.1 (200.62) | 980.8 (360.29) | 932.7 (263.27)

10. Secondary Outcome: Plasma Concentration of PF-04191834
Time Frame: Pre-dose and post-dose (1 to 3 hours) on Days 1, 8, 15, 29, 36, and 43
Population: Due to early termination of the study, only a subset of pharmacokinetic (PK) samples, from 10 out of 190 randomized participants, were selected for analysis. These 10 participants were selected based on treatment and treatment sequence.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- PF-04191834 600 mg BID: PF-04191834 600 mg BID administered either in Period 1 or Period 2
- PF-04191834 600 mg BID + Naproxen 500 mg BID: PF-04191834 600 mg BID plus naproxen 500 mg BID administered either in Period 1 or Period 2
Arm/Group | PF-04191834 600 mg BID | PF-04191834 600 mg BID + Naproxen 500 mg BID
Number analyzed (Participants) | 5 | 5
ng/mL
  Period 1 Day 1 Post-dose | 121.5 (7.7782) | 214.8 (280.61)
  Period 1 Day 8 Pre-dose | 623.5 (381.13) | 1155 (236.32)
  Period 1 Day 8 Post-dose | 511.0 (246.07) | 1117 (209.29)
  Period 1 Day 15 Pre-dose | 1007 (61.518) | 843.0 (509.31)
  Period 1 Day 15 Post-dose | 797.5 (171.83) | 736.0 (440.86)
  Period 2 Day 29 Post-dose | 122.1 (175.93) | 137.3 (67.458)
  Period 2 Day 36 Pre-dose | 581.2 (508.08) | 1141 (918.53)
  Period 2 Day 36 Post-dose | 550.4 (472.91) | 1154 (787.01)
  Period 2 Day 43 Pre-dose | 137.9 (191.11) | 1271 (847.11)
  Period 2 Day 43 Post-dose | 127.5 (177.46) | 1181 (918.53)

11. Secondary Outcome: Urinary Leukotriene E4 (LTE4) Levels
Description: LTE4 is a terminal metabolic product of arachidonic acid by 5-LO. Its synthesis is dependent upon the activity of 5-LO and it is eliminated through urinary clearance. Hence, the level of urinary LTE4 (uLTE4) excretion may be an indicator of endogenous 5-LO activity.
Time Frame: Day -7 (Visit 2) up to Day 43 (Visit 9 or End of Treatment Period 2)
Population: Since the study was terminated prematurely for a potential safety signal, and in light of the efficacy analysis, the pharmacodynamic (PD) assessment of uLTE4 was not performed and no data are reportable.
Arm/Group | PF-04191834 Followed by Placebo | Placebo Followed by PF-04191834 | PF-04191834 + Naproxen Followed by Naproxen | Naproxen Followed by PF-04191834 + Naproxen
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- PF-04191834: PF-04191834 600 mg BID administered either in Period 1 or Period 2
- Placebo: Placebo administered either in Period 1 or Period 2
- PF-04191834 + Naproxen: PF-04191834 600 mg BID plus naproxen 500 mg BID administered either in Period 1 or Period 2
- Naproxen: Naproxen 500 mg BID administered either in Period 1 or Period 2
Arm/Group | PF-04191834 | Placebo | PF-04191834 + Naproxen | Naproxen
Serious Adverse Events (participants affected / at risk) | 0/79 | 1/81 | 2/81 | 0/83
Other Adverse Events (participants affected / at risk) | 35/79 | 43/81 | 39/81 | 42/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04191834 (N=79) | Placebo (N=81) | PF-04191834 + Naproxen (N=81) | Naproxen (N=83)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04191834 (N=79) | Placebo (N=81) | PF-04191834 + Naproxen (N=81) | Naproxen (N=83)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Nodal arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Conjuctivitis (Eye disorders) | 1 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 3 | 0
Abnormal faeces (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 4 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 2 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 | 3
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 5 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0
Facial pain (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 1 | 1
Oedema peripheral (General disorders) | 1 | 1 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 2 | 1
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 2 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 4 | 1 | 2 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 5 | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Eye penetration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 1
ECG signs of myocardial ischaemia (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 2 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0
Heart sounds abnormal (Investigations) | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0 | 2
Arthritis (Metabolism and nutrition disorders) | 3 | 3 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 1 | 2
Bursitis (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 1
Headache (Nervous system disorders) | 6 | 5 | 5 | 8
Hemicephalalgia (Nervous system disorders) | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Mental impairment (Nervous system disorders) | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 1 | 1
Suicidal ideation (Nervous system disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Asteatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early due to increases in hepatic enzymes for which a relationship to study drug could not be excluded and that could alter the potential benefit-risk for participants continuing in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.